CLINICAL TRIAL: NCT05791019
Title: Efficacy of Paleolithic Diet in Control of Blood Level of Glucose in Type 2 DM Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nagy Nageh Abdo, Assistant lecturer, Assiut University
Other Study IDs: Paleolithic diet and T2DM
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: Paleolithic diet effect on patients — Efficacy of paleolithic diet in control of blood level of glucose in type 2 DM patients

SUMMARY:
Efficacy of paleolithic diet in control of blood glucose level in type 2 DM patients

DETAILED DESCRIPTION:
Diabetes mellitus has become one of the most common progressive chronic diseases in the world, with 422 million people affected worldwide. Approximately 95% of people currently diagnosed with diabetes have type 2 diabetes mellitus (T2DM). The disease is characterized by chronic hyperglycemia, which can impair pancreatic beta cell function and increase insulin resistance, deteriorating the metabolic condition and causing microvascular complications in the retina, kidney or peripheral nerves . Thus, glycemic control is essential for diabetes management, in order to avoid complications in organs and systems, which are related with high morbidity and mortality rates. Among T2DM causes are genetic and epigenetic elements interacting within a societal framework. The genetic predisposition for T2DM takes into account the increased risk of an individual to develop T2DM when there are other family members affected. On the other hand, epigenetic elements are those influenced by environmental factors, i. e., they can be reversible, and therefore manipulated, in order to treat the disease. Regardless of the causes, the main targets of the treatment are focused on decreasing insulin resistance and improving beta cell function and decrease the inflammatory process through diet, exercise and antihyperglycemic agents. Based on this, given the high prevalence of the disease and the significant benefits of its management, it is of clinical importance to determine the proper amount and type of carbohydrates in patients' diet, as they both may influence the glycemic index of a meal. Besides, some foods' intake induce a marked rise followed by a more or less rapid fall in blood glucose, while others produce a smaller peak along with a more gradual decline in plasma glucose. Currently, it is recommended for T2DM patients an intake of 26-44% of total daily energy from carbohydrates, preferably from high-quality sources, such as vegetables, whole fruits and legumes , which are rich in fiber. Most fibers, which are unabsorbed carbohydrates, are insoluble and increase stool weight. In contrast, starches are carbohydrates found in vegetables that are mostly broken down to sugars by digestive enzymes. Resistant starch, also found in vegetables and whole fruits, escapes digestion, being fermented in the intestine as well as dietary fiber. Although the quantity and the quality of carbohydrates in the diet influence blood glucose levels , influencing insulin secretion and gastric emptying, the most beneficial type, the ideal amount of dietary carbohydrates and the underlying mechanisms involved remain a matter of debate. Thus, this study was designed to systematically review the effects of the type and amount of dietary carbohydrates in studies involving T2DM , in order to clarify these aspects for improving T2DM management.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 DM, age less than 45 years old

Exclusion Criteria:

* type 1 DM infection bariatric surgery not follow diet regimine before study at least 6 month not on medication for weight reduction

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Newly diagnosed type 2 DM, age less than 45 years old, not less than 5 years of DM, not diagnosed to have type 1 DM, not having infection, not having history of bariatric surgery and not following deut regimen for weight reduction
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of paleolithic diet in control of blood glucose levels in type 2 DM patients | Baseline
  Controlling of glucose levels in blood by using specific dietary system and notifying the number of participants who achieve good results

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Abbas Said Muhammad El-Masry, Prof, Study Director — Assiut university hospitals
Locations (1):
- Nagy Nageh Abdo, Asyut, Egypt

REFERENCES:
- [Background] Kleiner A, Cum B, Pisciotta L, Cincione IR, Cogorno L, Prigione A, Tramacere A, Vignati A, Carmisciano L, Sukkar SG. Safety and Efficacy of Eucaloric Very Low-Carb Diet (EVLCD) in Type 1 Diabetes: A One-Year Real-Life Retrospective Experience. Nutrients. 2022 Aug 5;14(15):3208. doi: 10.3390/nu14153208. PMID 35956384